CLINICAL TRIAL: NCT00998803
Title: Surveillance of Influenza Virus Shedding and Immunologic Response in Immunocompromised Children and Young Adults
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FLUSRV
Record Dates: First submitted 2009-10-19; First posted 2009-10-21 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Influenza Virus
Keywords: Influenza virus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Nasopharyngeal swab collection is as follows: after tilting the tip of the patient's nose upward, a swab is inserted through the nostril along the floor of the nose into the nasopharynx. Then, the swab is gently rotated, removed and placed in its receptacle for delivery to the laboratory.
  * Respiratory specimens will be stored at 2-8ºC and processed within 24-48 hours of collection. Serum and whole blood for immune assays will be frozen at -20ºC or in liquid nitrogen until processed in batched assays.
  * All blood specimens will be sent to the laboratory for immunologic assays.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Immunocompromised participants: Immunocompromised (<= 21 years of age) due to cancer, receipt of stem cell transplant, human immunodeficiency virus (HIV) or Sickle cell disease

SUMMARY:
Influenza virus infections are a major cause of morbidity and mortality. The limited existing knowledge about the impact of influenza in immunocompromised patients suggests that they are at increased risk of influenza virus acquisition, of developing complications and of prolonged illness and viral shedding. However, some other data about the effect of antiviral agents on the infection course, and risk of resistance in immunocompromised children are lacking. The emergence of the pandemic H1N1 swine-origin influenza A virus has generated an additional need to study the epidemiology, clinical course and outcome of influenza infections in immunocompromised children. This study proposed to conduct a prospective observational clinical study to answer these questions.

DETAILED DESCRIPTION:
This study aims to do the following;

* To evaluate the frequency of influenza virus infections due to various subtypes in immunocompromised children and young adults at SJCRH
* To describe and compare the clinical course and outcome of pandemic H1N1 influenza infection with that due to other influenza virus subtypes in immunocompromised children and young adults.
* To evaluate the duration of influenza virus shedding in immunocompromised children and young adults.
* To evaluate the immunologic response to natural infection with various subtypes of influenza virus including the pandemic H1N1 influenza A virus.
* To evaluate the viral resistance to antiviral agents in relation to antiviral therapy.
* To compare accuracy of rapid methods for influenza A subtyping and for determination of antiviral resistance.

ELIGIBILITY:
Inclusion Criteria:

* Age <= 21 years of age at the time of entry into the study.
* Body weight of 13 kg or greater
* An immunosuppressed state due to cancer, sickle cell disease, HIV, or receipt of stem cell transplant
* Presentation with acute respiratory illness defined as recent onset of rhinorrhea, nasal and sinus congestion, pharyngitis, coryza, sinusitis, otitis media, dyspnea or shortness of breath, cough and/or a new radiographic pulmonary infiltrates.
* Proven influenza virus infection by virological testing of respiratory specimens using Polymerase Chain reaction (PCR) assay, direct antigen detection assay, or viral culture.

Exclusion Criteria:

* Inability or unwillingness of research participant or legal guardian to give written informed consent.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This is a prospective surveillance study that evaluates research participants who are ≤ 21 years of age and diagnosed at SJCRH with acute respiratory illness due to influenza virus confirmed by antigen detection, PCR or viral culture of clinical respiratory specimens.
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2009-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the frequency of influenza virus infections due to various subtypes in immunocompromised children and young adults at SJCRH | one year after enrollment

SECONDARY OUTCOMES:
To describe and compare the clinical course and outcome of pandemic H1N1 influenza virus infection with that due to other influenza virus subtypes in immunocompromised children and young adults. | one year after enrollment
To evaluate the duration of influenza viral shedding in immunocompromised children and young adults. | one year after enrollment
To evaluate the immunologic response to natural infection with various subtypes of influenza virus including the pandemic H1N1 virus. | one year after enrollment
To evaluate the viral resistance to antiviral agents in relation to antiviral therapy. | one year after enrollment
To compare accuracy of rapid methods for influenza A subtyping and for determination of antiviral resistance. | one year after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Hana Hakim, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St . Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org